CLINICAL TRIAL: NCT05050539
Title: Testing an Adaptive Implementation Strategy to Optimize Delivery of Obesity Prevention Practices in Early Care and Education Settings
Brief Title: Adaptive Implementation to Optimize Delivery of Obesity Prevention Practices in Early Care and Education Settings
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: Louisiana Tech University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: 262638
Record Dates: First submitted 2021-08-23; First posted 2021-09-20 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Obesity, Childhood; Nutrition Aspect of Cancer
MeSH Terms: conditions — Pediatric Obesity | interventions — Ultrasonic Waves

STUDY DESIGN:
Intervention Model Description: An enhanced non-responder trial design will be used to determine the effectiveness (Aim 1) and incremental cost-effectiveness (Aim 3) of an adaptive implementation strategy for WISE, while examining moderators and mediators of the strategy effect (Aim 2). In this trial, sites that do not respond to low-intensity strategies will be randomized to either (a) continue receiving low-intensity strategies or (b) receive high-intensity strategies. This design will determine the effect of an adaptive implementation strategy that adds high intensity versus one that continues with low intensity among non-responder sites.
Who Masked: Participant, Outcomes Assessor
Masking Description: Trained and field-reliable staff blinded to the study condition will collect data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Early Responders to Low Intensity (Active Comparator): Early responders will include those with targeted levels of fidelity by the October assessment. They will continue to receive low intensity implementation support (i.e., formal commitments, local champions, implementation blueprint, reminder cutting boards, task-focused implementation).
  Interventions: Behavioral: Low Intensity
- Non-Responders Continue Low Intensity (Active Comparator): This group will include those not achieving desired levels of fidelity by the October assessment who will be randomized to continue receiving low intensity implementation support (i.e., formal commitments, local champions, implementation blueprint, reminder cutting boards, task-focused implementation).
  Interventions: Behavioral: Low Intensity
- Non-Responders Increasing to High Intensity (Experimental): This group will include those not achieving desired levels of fidelity by the October assessment who will be randomized to have high intensity support added (low intensity + holistic individualized facilitation, tailored educational materials).
  Interventions: Behavioral: Low Intensity; Behavioral: High Intensity

INTERVENTIONS:
Behavioral: Low Intensity — 5 implementation strategies: formal commitments, local champions, implementation blueprint , remind educators (cutting board with WISE EBPs), task-focused facilitation.
Behavioral: High Intensity — Low intensity implementation strategies with the addition of holistic individualized facilitation and tailored educational materials.
  Arms: Non-Responders Increasing to High Intensity

SUMMARY:
"Together, We Inspire Smart Eating" (WISE) is an intervention that improves children's diets in ECE. WISE includes 4 key evidence-based practices (EBPs): (1) hands-on exposures to fruits and vegetables, (2) role modeling by educators, (3) positive feeding practices, and (4) a mascot associated with fruits and vegetables. Standard implementation approaches to WISE result in suboptimal implementation of WISE EBPs. Additional implementation strategies are needed to increase adoption and fidelity to EBPs.

To date, most studies have employed an "all-or-nothing" approach, comparing multifaceted strategies to control groups without implementation support. Thus, there is an urgent need for optimized strategies that tailor implementation support intensity to the unique challenges and limited resources of the ECE context. The overall objectives of this application are to determine the effectiveness and cost-effectiveness of an adaptive implementation approach to improve adoption of the EBPs of WISE while also examining implementation mechanisms. The central hypothesis is that the addition of high-intensity strategies at sites that do not respond to low-intensity strategies will improve implementation and health outcomes.

DETAILED DESCRIPTION:
In the US, 4 out of 10 children are overweight or obese by age, and few children between 2 and 5 years old meet dietary guidelines. Consuming a healthy diet (e.g., fiber, antioxidant-rich foods) and maintaining a healthy weight protect against cancer and cancer-related mortality. Arkansas and Louisiana are among the states with the highest obesity rates, lowest quality diets, and highest cancer rates in the US. Given that early life patterns track into adulthood, early interventions are needed to decrease cancer risk later in life. Importantly, studies in early care and education (ECE, i.e., childcare) found that 80% of dietary programs and 70% of programs focusing on health behaviors demonstrated positive effects. Thus, ECE is a promising cancer prevention setting. However, intervention implementation in ECE is a challenge.

""Together, We Inspire Smart Eating" (WISE) is an intervention that improves children's diets in ECE. WISE includes 4 key evidence-based practices (EBPs): (1) hands-on exposures to fruits and vegetables, (2) role modeling by educators, (3) positive feeding practices to support children's self-regulation, and (4) a mascot associated with fruits and vegetables. Prior work by the study team documented that standard implementation approaches to WISE (i.e., training and reminders only) result in suboptimal implementation of WISE EBPs. Additional implementation strategies are needed to increase adoption and fidelity to EBPs.

To date, few studies have compared implementation strategies to improve EBP uptake in ECE. Available studies have had a strong emphasis on policy, with results supporting the positive effect of multifaceted strategies. However, these studies often used an "all-or-nothing" approach, comparing costly multifaceted strategies to control groups with no implementation support. Knowledge is limited on the intensity of implementation strategies that are needed to yield success; some organizations may need more intense strategies than others. Thus, there is a critical need for optimized implementation strategies that tailor intensity (high vs. low) to the unique challenges and limited resources of ECE. Further, understanding how strategies work and for whom (i.e., implementation mechanisms) will advance implementation efforts in ECE.

The research team's foundational work (K01-DK110141) showed that a high-intensity implementation strategy package outperformed a standard implementation for WISE. However, it is likely not possible or necessary to provide a high-intensity strategy to all sites in wider dissemination. The proposed project will determine the optimal implementation intensity needed to improve the uptake of WISE EBPs in ECE. The overall objectives of this project are to determine the effectiveness and cost-effectiveness of an adaptive implementation approach to improve adoption of the WISE EBPs while also examining moderators and mediators of response to the strategies. The central hypothesis is that the addition of high-intensity strategies at sites that do not respond to low-intensity strategies will improve implementation and health outcomes compared to the continuation of low-intensity strategies. The research team's long-term goal is to increase EBP implementation in the ECE setting to improve health outcomes for children. Thus, the following specific aims are proposed:

Specific Aim 1. Determine the effectiveness of an adaptive implementation strategy that tailors the intensity of implementation support versus a low-intensity strategy. Using an enhanced non-responder trial, we will compare the effect of continuing low-intensity strategies vs. augmenting with high-intensity strategies to implement WISE. Low-intensity includes task-focused facilitation aimed at leaders; high intensity includes holistic, individualized facilitation aimed at educators. Non-responder sites (N =64) will be randomized to continue with the low-intensity strategies or to add high-intensity strategies. The hypothesis is that, on average, sites receiving high-intensity strategies will outperform sites continuing the low-intensity strategies on the primary outcome of intervention fidelity and on secondary implementation and child health outcomes.

Specific Aim 2. Examine moderators and mediators of implementation outcomes in a mixed-methods design. For moderation, the hypothesis is that sites with weaker organizational readiness and less experienced educators will require high intensity strategies to reach fidelity. For mediation, the expectation is that educators' perceptions of barriers, implementation climate, and implementation leadership will mediate the effect of the strategies on implementation outcomes. Using an explanatory, sequential design, qualitative data at purposively selected sites (N =20) will be collected to identify emergent moderators and mediators.

Specific Aim 3. Assess the incremental cost-effectiveness of the adaptive implementation strategy. In this aim, cost per unit of fidelity associated with the adaptive implementation strategy will be estimated based on a meaningful difference in the research team's previously published fidelity measure. Results will also determine the incremental cost-effectiveness of applying the adaptive strategy compared to continuing low-intensity strategies for improving child health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Recruited teachers at participating early care and education site in the following 4 geographic regions: (1) Central Arkansas, (2) Arkansas River Valley, (3) North, Central Louisiana, and (4) Southeast Louisiana.
* Participation in Child and Adult Care Food Program in the states' quality rating system
* Serving at least 15 children age 3 to 5
* Agreeing to participate in implementation activities and data collection in all 3- to 5-year-old classrooms
* Having no classrooms currently using WISE.

Exclusion Criteria:

* Having classrooms currently using WISE.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1850 (Estimated)
Dates: Start 2022-06-14 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Fidelity to WISE Evidence-Based Practices using the WISE fidelity observational measure | Through study completion, an average of 2 years
  Fidelity to the WISE Evidence-Based Practices at the classroom level measured with the the WISE fidelity observational measure.
  The measure includes 2 to 3 items per evidence-based practice (EBP) on a 1 (minimum) to 4 (maximum) scale to receive an average, continuous fidelity score with 4 representing the highest fidelity (i.e., higher scores reflect better fidelity). For each item, values are anchored to concrete, observable behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Taren M Swindle, Ph.D., Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No
After completion of the study, a database that includes de-identified participant information will be constructed, and this database will be accompanied by a detailed data dictionary that describes each variable by variable name, variable description, variable type (numeric, text, date), and acceptable variable ranges.

REFERENCES:
- [Derived] Swindle T, Rutledge JM, Selig JP, Painter J, Zhang D, Martin J, Johnson SL, Whiteside-Mansell L, Almirall D, Barnett-McElwee T, Curran GM. Obesity prevention practices in early care and education settings: an adaptive implementation trial. Implement Sci. 2022 Mar 18;17(1):25. doi: 10.1186/s13012-021-01185-1. PMID 35303894

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-23): https://cdn.clinicaltrials.gov/large-docs/39/NCT05050539/Prot_SAP_000.pdf